CLINICAL TRIAL: NCT06830148
Title: Effectiveness of Post-Procedural Manual Manipulation for Infant Ankyloglossia in Enhancing Breastfeeding and Reducing Revision Rates: a Prospective Randomized Trial
Brief Title: Post-Procedural Manual Manipulation for Infant Ankyloglossia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Earl H. Harley, Jr., MD, Chief of Pediatric Otolaryngology and Professor of Otolaryngology and Pediatrics, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00008313
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Ankyloglossia; Breastfeeding Support
Keywords: tongue tie; breastfeeding; exercises; infant; pediatric otolaryngology; frenotomy
MeSH Terms: conditions — Ankyloglossia; Breast Feeding; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Experimental): In the treatment group, parents will be instructed to perform postprocedural manipulation after the frenotomy.
  Interventions: Other: Post-frenotomy manual manipulation
- Control Group (No Intervention): In the control group, parents will not receive any instructions to perform "suck re-training" exercises or stretching following the procedure.

INTERVENTIONS:
Other: Post-frenotomy manual manipulation — Parents assigned to the treatment group will be instructed to perform post-frenotomy stretches and exercises four times daily, after every other feed, until the time of their postoperative visit 2-3 weeks later.
  Other Names: Post-procedural exercises
  Arms: Exercise Group

SUMMARY:
The goal of this randomized control trial is to determine the impact of post-frenotomy manual manipulation on revision rates and breastfeeding outcomes. We hypothesize that post-frenotomy manipulation will reduce the rate of sublingual frenulum regrowth, and subsequently frenotomy revision rates, thereby improving breastfeeding performance.

Infants with ankyloglossia undergoing frenotomy will be randomized into two groups: the intervention group (post-frenotomy manipulation) and the control group (no intervention). Parents in the intervention group will be instructed to perform tongue stretching and suck "re-training" exercises four times daily for 2-3 weeks, beginning 24 hours post-procedure. To monitor adherence and assess any complications, investigators will conduct a follow-up phone call one week after the procedure. Parents in the control group will not be instructed to perform any post-procedural manipulation. All participants will have a mandatory in-person follow-up 2-3 weeks postoperatively, during which breastfeeding outcomes and the need for frenotomy revision will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* infants less than 90 days old with ankyloglossia who undergo outpatient frenotomy using cold-steel scissors and will be exclusively or partially breastfed.

Exclusion Criteria:

* infants older than 90 days, those who will be exclusively bottle fed, infants who undergo concomitant lip tie release, those who undergo laser frenotomy, and infants who have previously undergone a frenotomy.
* infants with a gestational age of less than 36 weeks, those in the NICU or post-partum unit, infants who didn't receive the vitamin K injection, and those with congenital anomalies or medical conditions affecting breastfeeding

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants who are recommended to undergo repeat frenotomy | From enrollment to the 2-3 week postoperative visit
  Recommendations for frenotomy revision will be made by the principal investigator during the post-operative visit, which occurs 2-3 weeks following the procedure. This will include a physical examination to assess post-operative healing, along with an evaluation of the mother's breastfeeding outcomes.
Improvement in breastfeeding performance following post-procedural manual manipulation | From enrollment to the 2-3 week postoperative visit
  Pre- and post-operative maternal breastfeeding performance will be assessed using the LATCH score, a validated questionnaire that evaluates breastfeeding effectiveness. The pre-operative score will be administered during the initial consultation, while the post-operative score will be taken at the follow-up visit, 2-3 weeks after the procedure. The difference in scores will be analyzed to determine if there is an improvement in maternal breastfeeding outcomes.

SECONDARY OUTCOMES:
Compliance with post-frenotomy stretching and exercises | From enrollment to the 1 week postoperative phone call
  Parents assigned to the treatment group will receive a phone call one week postoperatively to assess their adherence to the treatment plan.

CONTACTS AND LOCATIONS:
Overall Officials: Earl H Harley, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- MedStar Georgetown University Hospital, Department of Otolaryngology-Head and Neck Surgery, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LeFort Y, Evans A, Livingstone V, Douglas P, Dahlquist N, Donnelly B, Leeper K, Harley E, Lappin S. Academy of Breastfeeding Medicine Position Statement on Ankyloglossia in Breastfeeding Dyads. Breastfeed Med. 2021 Apr;16(4):278-281. doi: 10.1089/bfm.2021.29179.ylf. No abstract available. PMID 33852342
- [Background] Messner AH, Walsh J, Rosenfeld RM, Schwartz SR, Ishman SL, Baldassari C, Brietzke SE, Darrow DH, Goldstein N, Levi J, Meyer AK, Parikh S, Simons JP, Wohl DL, Lambie E, Satterfield L. Clinical Consensus Statement: Ankyloglossia in Children. Otolaryngol Head Neck Surg. 2020 May;162(5):597-611. doi: 10.1177/0194599820915457. Epub 2020 Apr 14. PMID 32283998